CLINICAL TRIAL: NCT05046509
Title: The Clinical Manifestations of SARS-Cov-2 Disease; Not Only Pulmonary
Brief Title: The Clinical Manifestations of the Severe Acute Respiratory Syndrome, Coronavirus 2( SARS-Cov-2 ); Not Only Pulmonary
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad eldin arafa Aly, Allergist and Immunologist, Assiut University
Other Study IDs: 17101489
Record Dates: First submitted 2021-09-03; First posted 2021-09-16 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID_Patients: * Patients have been confirmed diagnosed with Covid-19 disease by PCR
  * Patients aged 18 years and above

SUMMARY:
A prospective observational study to identify different extrapulmonary clinical manifestations of SARS-CoV-2 and its correlations with the disease severity grades.

DETAILED DESCRIPTION:
The current research in this area was retrospective trials; this study is a prospective one. Investigators will perform the extensive recording of extrapulmonary manifestations in adult patients of SARS-CoV-2 and their correlations with the disease severity grades.

Type of the study: a prospective observational study

Study Setting:

Data will be collected from outpatients and inpatients files and a questionnaire.

Sample Size Calculation:

Depending on the average monthly (40-50 cases) and type of the study :

-Investigators will use Steven K. Thompson equation 13 to calculate the size from the next formula

Population size =(752) Sample size = (414) Level of confidence: ( 95%) Error proportion: (0.05) Probability :(20 %) Study power: (80 %)

ELIGIBILITY:
Inclusion Criteria:

* Patients have been confirmed diagnosed with Covid-19 disease by PCR
* Patients aged 18 years and above

Exclusion Criteria:

* Patients aged below 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected from outpatients and inpatients files.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Number of participants who has one or more of the following extrapulmonary clinical manifestations of SARS-CoV-2 . | one year
  Cardiovascular :
  * Coronary Artery Disease
  * Infarction (type 2)
  * Myocarditis
  * Arrhythmia
  * Cardiogenic shock
  * Heart failure
  Gastrointestinal :
  * Anorexia
  * Diarrhea
  * Bleeding
  * Digestive symptoms
  * Abnormal liver tests
  Neurological :
  * Headache
  * Impaired consciousness
  * acute ischemic stroke
  * Ataxia
  * Dizziness
  * Seizure
  * Taste impairment
  * Smell impairment
  * Vision impairment
  * Viral encephalitis
  * Depression
  Endocrinal:
  * Hypoglycemia
  * Ketoacidosis
  * Hyperglycemia
  * Thyrotoxicosis
  * Secondary Adrenal Insufficiency
  Hematological:
  * Leukocytosis
  * Leukopenia
  * Thrombocytopenia
  * Anemia
  * Lymphocytosis
  * D-dimer
  * Lactate dehydrogenase
  * Ferritin
  Renal :
  * Albuminuria
  * Hematuria
  * Blood urea nitrogen
  * Acute kidney injury
  Ophthalmologic :
  -Conjunctivitis
  Dermatologic :
  * Papulovesicular rash
  * Rosacea
  * Dryness
  * Erythema
  * Urticaria
  * Maculopapular exanthem morbilliform

SECONDARY OUTCOMES:
The correlations between the number of participants who has extrapulmonary manifestations and the severity grade of SARS-CoV-2. | one year
  These correlations between the number of participants who has one or more of extrapulmonary manifestations and the severity of SARS-CoV-2, will be measured.
  There are four severity grades of SARS-CoV-2 according to WHO classifications (mild, moderate, severe and critical)

CONTACTS AND LOCATIONS:
Overall Officials: Emad arafa, Msc, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xiao F, Tang M, Zheng X, Liu Y, Li X, Shan H. Evidence for Gastrointestinal Infection of SARS-CoV-2. Gastroenterology. 2020 May;158(6):1831-1833.e3. doi: 10.1053/j.gastro.2020.02.055. Epub 2020 Mar 3. No abstract available. PMID 32142773
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Zhu L, She ZG, Cheng X, Qin JJ, Zhang XJ, Cai J, Lei F, Wang H, Xie J, Wang W, Li H, Zhang P, Song X, Chen X, Xiang M, Zhang C, Bai L, Xiang D, Chen MM, Liu Y, Yan Y, Liu M, Mao W, Zou J, Liu L, Chen G, Luo P, Xiao B, Zhang C, Zhang Z, Lu Z, Wang J, Lu H, Xia X, Wang D, Liao X, Peng G, Ye P, Yang J, Yuan Y, Huang X, Guo J, Zhang BH, Li H. Association of Blood Glucose Control and Outcomes in Patients with COVID-19 and Pre-existing Type 2 Diabetes. Cell Metab. 2020 Jun 2;31(6):1068-1077.e3. doi: 10.1016/j.cmet.2020.04.021. Epub 2020 May 1. PMID 32369736
- [Background] Li J, Gong X, Wang Z, Chen R, Li T, Zeng D, Li M. Clinical features of familial clustering in patients infected with 2019 novel coronavirus in Wuhan, China. Virus Res. 2020 Sep;286:198043. doi: 10.1016/j.virusres.2020.198043. Epub 2020 Jun 2. PMID 32502551
- [Background] Perico L, Benigni A, Remuzzi G. Should COVID-19 Concern Nephrologists? Why and to What Extent? The Emerging Impasse of Angiotensin Blockade. Nephron. 2020;144(5):213-221. doi: 10.1159/000507305. Epub 2020 Mar 23. PMID 32203970
- [Background] Patel S, Rauf A, Khan H, Abu-Izneid T. Renin-angiotensin-aldosterone (RAAS): The ubiquitous system for homeostasis and pathologies. Biomed Pharmacother. 2017 Oct;94:317-325. doi: 10.1016/j.biopha.2017.07.091. Epub 2017 Jul 31. PMID 28772209
- [Background] Lanza K, Perez LG, Costa LB, Cordeiro TM, Palmeira VA, Ribeiro VT, Simoes E Silva AC. Covid-19: the renin-angiotensin system imbalance hypothesis. Clin Sci (Lond). 2020 Jun 12;134(11):1259-1264. doi: 10.1042/CS20200492. PMID 32507883
- [Background] Gembardt F, Sterner-Kock A, Imboden H, Spalteholz M, Reibitz F, Schultheiss HP, Siems WE, Walther T. Organ-specific distribution of ACE2 mRNA and correlating peptidase activity in rodents. Peptides. 2005 Jul;26(7):1270-7. doi: 10.1016/j.peptides.2005.01.009. Epub 2005 Feb 16. PMID 15949646
- [Background] Xu H, Zhong L, Deng J, Peng J, Dan H, Zeng X, Li T, Chen Q. High expression of ACE2 receptor of 2019-nCoV on the epithelial cells of oral mucosa. Int J Oral Sci. 2020 Feb 24;12(1):8. doi: 10.1038/s41368-020-0074-x. PMID 32094336
- [Background] Zou X, Chen K, Zou J, Han P, Hao J, Han Z. Single-cell RNA-seq data analysis on the receptor ACE2 expression reveals the potential risk of different human organs vulnerable to 2019-nCoV infection. Front Med. 2020 Apr;14(2):185-192. doi: 10.1007/s11684-020-0754-0. Epub 2020 Mar 12. PMID 32170560
- [Background] Martinez-Rojas MA, Vega-Vega O, Bobadilla NA. Is the kidney a target of SARS-CoV-2? Am J Physiol Renal Physiol. 2020 Jun 1;318(6):F1454-F1462. doi: 10.1152/ajprenal.00160.2020. Epub 2020 May 15. PMID 32412303
- [Background] Carsetti R, Quintarelli C, Quinti I, Piano Mortari E, Zumla A, Ippolito G, Locatelli F. The immune system of children: the key to understanding SARS-CoV-2 susceptibility? Lancet Child Adolesc Health. 2020 Jun;4(6):414-416. doi: 10.1016/S2352-4642(20)30135-8. Epub 2020 May 6. No abstract available. PMID 32458804
- [Background] [13] Steven K Thomson sampling 2012 third edition P 59-60
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Hirsch JS, Ng JH, Ross DW, Sharma P, Shah HH, Barnett RL, Hazzan AD, Fishbane S, Jhaveri KD; Northwell COVID-19 Research Consortium; Northwell Nephrology COVID-19 Research Consortium. Acute kidney injury in patients hospitalized with COVID-19. Kidney Int. 2020 Jul;98(1):209-218. doi: 10.1016/j.kint.2020.05.006. Epub 2020 May 16. PMID 32416116
- [Background] Wu P, Duan F, Luo C, Liu Q, Qu X, Liang L, Wu K. Characteristics of Ocular Findings of Patients With Coronavirus Disease 2019 (COVID-19) in Hubei Province, China. JAMA Ophthalmol. 2020 May 1;138(5):575-578. doi: 10.1001/jamaophthalmol.2020.1291. PMID 32232433
- [Background] Galvan Casas C, Catala A, Carretero Hernandez G, Rodriguez-Jimenez P, Fernandez-Nieto D, Rodriguez-Villa Lario A, Navarro Fernandez I, Ruiz-Villaverde R, Falkenhain-Lopez D, Llamas Velasco M, Garcia-Gavin J, Baniandres O, Gonzalez-Cruz C, Morillas-Lahuerta V, Cubiro X, Figueras Nart I, Selda-Enriquez G, Romani J, Fusta-Novell X, Melian-Olivera A, Roncero Riesco M, Burgos-Blasco P, Sola Ortigosa J, Feito Rodriguez M, Garcia-Doval I. Classification of the cutaneous manifestations of COVID-19: a rapid prospective nationwide consensus study in Spain with 375 cases. Br J Dermatol. 2020 Jul;183(1):71-77. doi: 10.1111/bjd.19163. Epub 2020 Jun 10. PMID 32348545